CLINICAL TRIAL: NCT02816905
Title: Ocular-hypertensive Response to Topical Steroids in Children After Bilateral Strabismus Surgery (Topical Rimexolone Versus Topical Dexamethasone and Topical Fluorometholone)
Brief Title: Ocular-hypertensive Response to Topical Steroids in Children After Bilateral Strabismus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Tawfik Al Hanaineh, Doctor Abeer Tawfik Farhan Al Hanaineh, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Abeer Al Hanaineh
Record Dates: First submitted 2016-06-26; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Intraocular Pressure
Keywords: intraocular pressure; topical steroids; strabismus
MeSH Terms: conditions — Strabismus | interventions — Dexamethasone; Steroids; Fluorometholone; rimexolone

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Group A (Active Comparator): 20 eyes that received topical 0.1% Dexamethasone 4 times per day for 2 weeks after surgery. And topical Moxifloxacin 4 times per day for 2 weeks after surgery.
  Interventions: Drug: 0.1 % Dexamethasone
- Group B (Active Comparator): 20 eyes that received topical 0.1 % Fluorometholone 4 times per day for 2 weeks after surgery. And topical Moxifloxacin 4 times per day for 2 weeks after surgery.
  Interventions: Drug: 0.1% Fluorometholone
- Group C (Active Comparator): 40 eyes that received topical 1% Rimexolone 4 times per day for 2 weeks after surgery. And topical Moxifloxacin 4 times per day for 2 weeks after surgery.
  Interventions: Drug: 1% Rimexolone

INTERVENTIONS:
Drug: 0.1 % Dexamethasone — 20 eyes are randomized to receive topical 0.1% Dexamethasone four times per day for 2 weeks.
  Other Names: Topical steroid
  Arms: Group A
Drug: 0.1% Fluorometholone — 20 eyes are randomized to receive topical 0.1% Fluorometholone four times per day for 2 weeks.
  Other Names: Topical steroid
  Arms: Group B
Drug: 1% Rimexolone — 40 eyes are randomized to receive topical 1% Rimexolone four times per day for 2 weeks. 20 of these eyes were the contralateral eyes of the patients who received 0.1% Dexamethasone in their first eye. The other 20 eyes were the contralateral eyes of the patients who received 0.1% Fluorometholone in their first eye
  Other Names: Topical steroid
  Arms: Group C

SUMMARY:
This study aims to compare the effects of topical (Rimexolone versus Dexamethasone) on the IOP in children under 13 years of age who underwent bilateral strabismus surgery, and to compare the effects of topical (Rimexolone versus Fluorometholone) on the IOP in the children under 13 years of age who underwent bilateral strabismus surgery.

DETAILED DESCRIPTION:
Children under the age of 13 years undergoing bilateral strabismus surgery in Cairo University Hospitals (Cairo University Specialized Pediatric Hospital and Kasr Al Ainy Hospital). will be randomized using simple randomization method, computer software for randomization, into two equal groups:

* First group: One eye is randomized to receive topical 0.1% Dexamethasone, whereas the fellow eye will receive topical 1% Rimexolone four times per day for 2 weeks.
* Second group: One eye is randomized to receive topical 0.1% Fluorometholone, whereas the fellow eye will receive topical 1% Rimexolone four times per day for 2 weeks.

IOP will be measured on the day before operation using the Tono-Pen®. Three reliable measurements will be obtained from each eye and the mean will be taken.

IOP will be measured at postoperative weeks 1, 2, 3, 4 and 6 using the Tono-Pen®.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than 13 years of age.
* Children who underwent bilateral recession strabismus surgeries.
* Preoperative IOP of 21.00 mmHg or less, with a cup-disc ratio of 0.3 or less.
* The absence of systemic disease and ocular disease (apart from strabismus) in both eyes.
* Children who can comply with the IOP measurements using the Tono-Pen®, as no type of anesthesia will be used, except for the topical anesthesia.

Exclusion Criteria:

* Patients that are 13 years of age or older.
* Children who need resection muscle surgeries, surgeries for the vertical, or the oblique muscles.
* Preoperative IOP of more than 21.00 mmHg, or a cup-disc ratio of more than 0.3
* Family history of glaucoma or high myopia.
* A history of steroid usage in the past year.
* Failure to comply with IOP measurements or the follow-up schedule.

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measuring the rise in intraocular pressure using the Tono-Pen® after topical steroids are used in children under 12 years of age, who underwent bilateral strabismus surgery | IOP will be followed up for 6 weeks after initial use
  Measuring the rise in intraocular pressure using the Tono-Pen® after topical steroid use in children. IOP will be measured at postoperative weeks 1, 2, 3, 4 and 6. And will be compared with pre-operative values.

CONTACTS AND LOCATIONS:
Overall Officials: Omar M. El Shafie El Zawahry, PhD, Study Chair — Cairo University Hospital- Department of Ophthalmology
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided